CLINICAL TRIAL: NCT01108029
Title: Study of Memantine to Treat Gait Disorders And Attention Deficit In Parkinson's Disease: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Monocentric Trial
Brief Title: Study of Memantine for Gait Disorders And Attention Deficit In Parkinson's Disease
Acronym: FOGG-I
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008-008210-38; 2008_02/0841 (Other: sponsor)
Record Dates: First submitted 2009-07-20; First posted 2010-04-21 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2009-07

CONDITIONS: Parkinson's Disease; Gait Disorders, Neurologic
Keywords: Parkinson's disease; Freezing of Gait; Memantine; NMDA receptor; glutamate; No Dementia
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- memantine (Active Comparator): memantine 20 mg/day (2 tablets 1 time a day in the morning)
  Interventions: Drug: memantine
- placebo (Placebo Comparator): 2 tablets (1 time a day in the morning) during 3 months
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: memantine — 2 tablets of 10 mg of memantine 1 time a day in the morning
  Other Names: EBIXA
  Arms: memantine
Drug: placebo — 2 tablets of placebo 1 time a day in the morning
  Arms: placebo

SUMMARY:
Along with cognitive and psychobehavioural disorders, gait disorders represent a major problem in the treatment of advanced Parkinson's disease (PD). PD can be considered to be a hyperglutamatergic disease because dopaminergic depletion induces hyperactivity of the subthalamic nucleus (STN) and the internal pallidum (GPi), with glutamatergic hyperactivity of the STN's efferent pathway, i.e., the subthalamopallidal, subthalamonigral and subthalamo-entopeduncular pathways (projecting to the pedunculopontine nucleus (PPN)). Excess glutamate in the PPN has also been observed in the 6-OHDA rat model of PD. Reduction of this glutamatergic hyperactivity within the PPN via the systemic or intra-peduncular administration of glutamate antagonists improves akinesia in drug-induced murine and primate models of PD, via the NMDA and AMPA receptors. High doses of memantine (10 mg/kg) improve locomotion in reserpine- and alpha-methyl-p-tyrosine-treated rats. In humans, the PPN may play a key role in gait, posture control, axial rigidity and attention. It is also involved in the gating of sensory information involved in the startle reflex, which can be studied via prepulse inhibition (PPI) of the blink reflex. At present, two uncompetitive NMDA receptor antagonists are approved for use in humans: amantadine and memantine. Reviews of the recent literature on these drugs have identified no published studies specifically on severe gait and attention disorders in PD. Memantine is a partial blocker of open NMDA channels. The value of memantine relates to the fact that it decreases excessive glutamatergic transmission by lowering the synaptic noise due to excessive activation of NMDA receptors. In this double-blind study, the investigators shall seek to demonstrate the presence or absence of an effect of memantine on gait and attention disorders. In order to study the interaction between glutamatergic hyperactivity and the dopaminergic system, the investigators shall study the phenomena both in the absence of L-dopa and following acute administration of the latter. Twenty eight volunteer, non-demented, late-stage PD patients displaying severe gait disorders will receive memantine (20 mg/day) or placebo for 3 months. The investigators expect to see a reduction in gait and attention disorders, together with an improvement in the blink reflex with PPI under memantine. This pilot study could subsequently be turned into a double-blind, placebo-controlled multicenter study.

DETAILED DESCRIPTION:
Overall study duration: 2 years. Planned inclusion period: 12 months. Study duration for individual patients: 4 months and 2 weeks(2 weeks between screening and randomization, 3 months of double-blind treatment and then a 4-week wash-out period).

Primary objective (V1 and V4):

To assess efficacy of memantine treatment on severe gait disorders assessed on stride length by gait analysis with an optoelectronic system (VICON®) in patients with advanced Parkinson's disease under subthalamic stimulation

Additional Efficacy Endpoints (V1 and V4):

* Kinematic and Kinetic parameters (stride length, stride time, velocity, and cadence) of the gait initiation and the stabilized gait using the optoelectronic system (VICON®)
* Gait and motor symptoms: the "Freezing Of Gait trajectory", the UPDRS scores (part III), the dyskinesia rating scale,
* Axial rigidity : measured by passive flexion on isokinetic dynamometer (Cybex 6000)
* Axial strength : measured by active flexion on isokinetic dynamometer (Cybex 6000)
* Attention: simple and complex reactions times
* The inhibition of the presynaptic dopamine transporter by memantine was assessed by the mean DAT density of the bilateral striatum (putamen and caudate nuclei) using [99mTc]TRODAT-1 SPECT

Safety and Tolerability Endpoints (V1, V2, V3 and V4):

* Drowsiness: Epworth and Parkinson's disease Sleep Scales
* Apathy Lille Apathy Rating Scale
* Depression : MADRS,
* Pharmacokinetic properties of memantine were analyzed by the lowest plasmatic concentrations of memantine before the morning intake of the blinded treatment at 7:00 h, during the steady state after 3 months (blind secondary analyse).
* Safety : Recording of all serious and non serious adverse events reported by the patients, electrocardiogram, blood pressure and biological analyzes (blood counts, ionogram, urea, creatinemia, transaminases, alkaline phosphatase, bilirubinemia, gamma GT, magnesium)
* Tolerability Number of subjects (%) who discontinue the study Number of subjects (%) who discontinue the study due to AEs Safety Measures AE incidence Safety laboratory values Vital signs Blood pressure monitoring ECG Physical and neurological examination

Study Design

Monocentric study: 12-week double blind, placebo-controlled phase. After being found eligible to participate in the study, subjects will be allocated in a 1:1 ratio into one of the following two treatment groups based on a randomization scheme with blocks stratified:

one memantine

1. st week: 5 mg per day in the morning
2. nd week: 10 mg per day in the morning
3. rd week: 15 mg per day in the morning
4. th week: 20 mg per day in the morning

one placebo during 3 months same as memantine

Schedule: 5 visits : screening (V0), randomization (V1, 15 days after V0), (V2) visit after 1 months, (V3) visit after 2 months and termination (V4, 3 months after randomization)

Patients : 28 subjects with Parkinson's disease duration of more than 5 years, without dementia (Mattis Dementia Rating Scale ≥ 130, MMSE ≥ 27 and DSM IV), without major depression (MADRS < 18) who have severe gait disorders including freezing of gait (defined by an answer 2 or 3 at the 3rd question of the autoquestionnaire of Giladi: Do your gait disorders impede your daily living activities and your independence: answer: yes, moderately or severely. But the patient requires no physical assistance to walk) despite an optimal dopaminergic treatment and optimal and stable subthalamic stimulation parameters. No additional therapy will be permitted during the study.

Centre : LILLE :

Department of Neurology, University Hospital of Lille : Pr L. Defebvre, Pr K. Dujardin, Dr D. Devos, Pr Destee, Mme Delliaux. Dr A Kreisler, Dr C Simonin, Dr C. Moreau, Dr A. Delval Department of Pharmacology, Faculté de Médecine, Lille II.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease of more than 5 years
* Subthalamic nucleus stimulation
* Gait disorders impeding moderately to severely the activities of daily living
* gait disorders including freezing of gait
* able to walk without physical assistance

Exclusion Criteria:

* Dementia (MMSE < 27 et score de Mattis < 130)
* Requiring dopatherapy modification
* Requiring subthalamic stimulation parameters adaptation
* Psychiatric disorders: hallucinations, unstable thymic disorders, psychosis)
* Cardiac disorders: dysrhythmia or unstable arterial hypertension
* Unstable or severe medical illness
* intolerance or contraindication to memantine

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-10; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
stride length by gait analysis with an optoelectronic system (VICON®) | 3 months of treatment

SECONDARY OUTCOMES:
Kinematic and Kinetic parameters (stride length, stride time, velocity, cadence and variability of these parameters) of the gait initiation and the stabilised gait using the optoelectronic system (VICON®) | 3 months
Gait and motor symptoms: the "Freezing Of Gait trajectory",the UPDRS motor score (part III), the dyskinesia rating scale, | 3 months
Attention: simple and complex reactions times | 3 months
hypertonia of axial flexor and extensor | 3 months
  hypertonia of axial flexor and extensor measured on mean and total work at 30°/s (Joules) by passive flexion and extension on isokinetic dynamometer (Cybex 6000)
Drowsiness: Epworth and Parkinson's disease Sleep Scales | 3 months
Apathy Lille Apathy Rating Scale | 3 months
Depression: MADRS | 3 months
Safety and Tolerability Endpoints | 3 months
  * Safety : Recording of all serious and non serious adverse events reported by the patients, electrocardiogram, blood pressure and biological analyzes (blood counts, ionogramme, urea, creatinemia, transaminases, alkaline phosphatase, bilirubinemia, gamma GT, magnesium)
  * Tolerability Number of subjects (%) who discontinue the study Number of subjects (%) who discontinue the study due to AEs Safety Measures AE incidence Safety laboratory values Vital signs Blood pressure monitoring ECG Physical and neurological examination
strength of axial flexor and extensor | 3 months
  strength of axial flexor and extensor measured on mean and total work of 3 repetitions at 30°/s (Joules) and of 5 repetitions at 120°/s (Joules) by active flexion and extension on isokinetic dynamometer
DaT scan | 3 months
  The inhibition of the presynaptic dopamine transporter by memantine was assessed by the mean DAT density of the bilateral striatum (putamen and caudate nuclei) using [99mTc]TRODAT-1 SPECT before and after 3 months of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: David Devos, MD, PhD, Principal Investigator — Department of Neurology, University Hospital of Lille
Locations (1):
- Devos, Lille, France

REFERENCES:
- [Derived] Moreau C, Delval A, Tiffreau V, Defebvre L, Dujardin K, Duhamel A, Petyt G, Hossein-Foucher C, Blum D, Sablonniere B, Schraen S, Allorge D, Destee A, Bordet R, Devos D. Memantine for axial signs in Parkinson's disease: a randomised, double-blind, placebo-controlled pilot study. J Neurol Neurosurg Psychiatry. 2013 May;84(5):552-5. doi: 10.1136/jnnp-2012-303182. Epub 2012 Oct 16. PMID 23077087